CLINICAL TRIAL: NCT04940884
Title: The Effects of Exercise Intervention on Health-related Physical Fitness and Circulating microRNA in the Community Senior Residents
Brief Title: Supervised Exercise Training Effects on Older Community Dwellers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: 201602058A3C502
Record Dates: First submitted 2021-06-14; First posted 2021-06-28 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Aging
Keywords: aerobic exercise; physical fitness; body compositions; micro rna

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised exercise training (Experimental): Pre- and Post- exercise training effects. Part of the participants were randomly assigned to underwent additional 24 sessions of supervised exercise training (SET) and the remaining participants follow the above instruction without additional supervised exercise training. After the 24 sessions of SET, they were then followed a 16-week of follow-up of their daily activities without additional exercise training.
  Interventions: Behavioral: Supervised exercise training; Behavioral: Aerobic exercise training
- home exercise training (Active Comparator): All included subjects were instructed to walk>=8000 steps per day (stp/d), which was recorded by wrist-worm smart watches
  Interventions: Behavioral: Aerobic exercise training

INTERVENTIONS:
Behavioral: Supervised exercise training — SET Participants underwent 24 sessions of moderate-intensity exercise training (MICT) at 70% maximum predicted heart rate for 30 min in each session
  Arms: Supervised exercise training
Behavioral: Aerobic exercise training — All recruited subjects were instructed to walk >=8000 steps per day in the community. Part of the participants were randomly assigned to underwent additional 24 sessions of supervised aerobic exercise training (SET) with the intensity at 70% of maximum predicted heart rate and the remaining participants follow the above home exercise training (HET) instruction without additional supervised exercise training.

SUMMARY:
Altered circulating microRNA (miRNA) after physical activity reflects exercise effects on muscle performance and cardiorespiratory fitness. The present work was designed to highlight associations between exercise-induced physical fitness miRNAs in community-indwelling elderly adults. Baseline clinical information was assessed for community-indwelling individuals, long-term followed by our community medicine research center, aged >=55 years near our hospital. Among them, participants were randomly assigned to the supervised exercise training (SET) and home exercise training (HET) groups. All included subjects were instructed to walk>=8000 steps per day (stp/d), which was recorded by wrist-worm smart watches. SET Participants underwent 24 sessions of moderate-intensity exercise training (MICT) at 70% maximum predicted heart rate for 30 min in each session. HET participants underwent walking activities as the above instruction. Movement analysis and body composition measurements were used to assess physical fitness at baseline and 8 as well as 24 weeks after recruitment. MiRNAs (miR-21, miR-126, miR-146a, and miR-222) were also examined at the above time point. SET participants took significantly more steps per day and had greater chance to walk>=8000 stp/d in the community compared to the SET participants during follow-up. Prominent beneficial effects on physical fitness, including cardiorespiratory fitness, flexibility, lower extremity muscle strength, and body composition, were noticed during and 16 weeks after stopping SET. Increased miR146a and miR-126 expressions reflecting increased anti-inflammatory response and enhanced angiogenesis, respectively after 8 weeks of SET. However, inhibited skeletal as well as cardiac muscle catabolism respectively reflecting in the increased miR-21 and miR-222 were also identified in the present work. These observations may clarify short-term SET effects on lifestyle in community inhabitants and how sensitive of miRNAs to exercise-induced physiological adaptations.

DETAILED DESCRIPTION:
Design The Institutional Review Board of a tertiary care hospital approved the study (IRB No.: 201602058A3C502 and NCT04839796). A randomized controlled trial with assessor and subject blinded study for effects of exercise regimens on ageing persons was performed from May to November 2021. All subjects provided informed consent after understanding the experimental procedures. Participants were then randomly allocated to undergo 30 min of supervised exercise training (SET) at moderate-intensity continuous training (MICT) for 24 sessions in the hospital or home exercise training (HET) groups using a computer-generated, concealed allocation schedule. Data were collected by a blinded assessor prior to randomization and after completing the exercise training.

Participants Community-indwelling individuals with age>=55 years, who lived adjacent to a community hospital were surveyed. Elderly adults with mini-mental state examination (MMSE) score > 24 and negative lumbar spine as well as lower extremity degenerative joint disorder were recruited. Those who had unstable clinical presentations mentioned in our previous studies, or sarcopenia, diagnosed based on the recommendation of the Asian Working Group for Sarcopenia, were not candidates of the study. We also excluded individuals with absolute contraindications for aerobic activities, suggested by the American College of Sports Medicine (ACSM). The baseline physical component score (PCS) and mental component scores (MCS) in the Medical Outcomes Study Short Form 36 (SF-36) were used to assess the quality of life (QoL) and were re-evaluated 24 weeks after the recruitment. Baseline demographic characteristics and clinical information of included participants were carefully recorded.

Exercise Training All subjects were instructed to wear a smart watch (WDI08, WisDat Inc., Taichung, Taiwan) and to take at least 8000 steps per day (stp/d). In addition to 8000 stp/d, the SET participants underwent 24 sessions of supervised MICT (70% of maximum predicted HR) for 30-min on a bicycle ergometer (Ergoselect 150P, ergoline GmbH, Bitz, Germany) in our hospital during an 8-week period. All subjects were reminded to take >=8000 stp/d every week during the first 8-week after recruitment by phone call and app. After completing the MICT, SET participants were instructed to take >=8000 stp/d for another 16 weeks. HET participants were instructed to take 8000 stp/d over the 24-week follow-up period. During the latter 16-week, the instruction of taking>=8000 stp/d was not reminded in all subjects. The exercise training was terminated when the subject had symptoms/signs during exercise according to the ACSM guideline.20 Measurement of physical fitness The wrist-worn smart watch (WDI08, Wisdat Inc., Taichung, Taiwan) recorded the every-day step count and energy expenditure in each subject, and the average number of steps and energy expenditure (Kcal) per day in a week represented the mean every day steps and energy expenditure of a week in community during the 24-week follow-up period.

The calf circumference (Calf_circ) was obtained by averaging the greatest Calf_circ in bilateral legs. Intelligent movement analysis (eFitHealth, uCare Medical Electronics, Co. Ltd., Miaoli, Taiwan) using interactive voices and 3D depth image guides to assess 2-min step number, 5-time sit-to-stand duration, and chair sit-and-reach distance (Supplementary Data 1). Each of the above test was used to estimate VO2max (eV O2max), lower extremity muscle strength, and flexibility, respectively.21 Body composition, including total body water (TBW), mineral portion, protein amount (Prot), lean body mass (LBM), skeletal muscle mass (SKM), body fat mass (BFM), and basal metabolic rate (BMR) were measured by multiple frequency bioimpedance analysis (Inbody 720, Inbody Co., Ltd., CA, USA). The above measurements were documented before, 8-week after, and 24-week after initial visit.

RNA extraction Blood sampling of 10 ml whole blood from each subject at the recruitment, 8-week, and 24-week from the initial visit was placed in a tube containing 3.2% sodium citrate. Samples were then centrifuged at 360xg for 15 min, which supernatant was further centrifuged at 2400xg for 20 min at room temperature of 25 ℃ to keep plasma platelet count less than 2.5×10^8/ml. Processed plasma of 400 microL was placed in a 2mL eppendorf (Eppendorf corp. Hamburg, Germany) to mix with 1200 microL TRIzol (ThermoFisher Scientific Inc., Waltham, MA, USA) and 5 microL miR-39 (5x10^-15 mol/microL), exogenous control, of C. elegans as well as 2 microg (10 microg/mL in plasma) yeast RNA (Invitrogen, Carlsbad, CA, USA) for 15 min at room temperature. Another 320 microL chloroform was added and placed at room temperature for 5 min. The specimen was centrifuged at 12000 xg for 15 min at 4 ℃ and 300 microL colorless fluid layer was aspirated to mix with 900 microL iced 100% ethanol overnight at -80 ℃. The prepared specimen was placed into the Direct-zol column (Direct-zol RNA Miniprep, Zymo Research corp., Irvine, CA, USA) and was then centrifuged at 12000 xg for 30 sec. The column was then transferred to a new collection tube and was centrifuged at 12000 xg for 30 sec after mixing with 400 microL RNA wash buffer. DNase I reaction mix of 80 microL (DNase I enzyme 5 microL+DNA digestion buffer 75 microL) was added to the tube after discarding the RNA wash buffer and was incubated at room temperature for 15 min. Additional 400 microL pre-wash buffer was introduced into the tube and was centrifuged at 12000 xg for 30 sec. The column was then transferred into a new 1.5 mL RNase-free tube and was treated with 80 microL nuclease-free water at room temperature for 2min. The prepared sample was centrifuged at 12000 xg for 2 min to elute RNA solution.

Quantification of plasma microRNA levels miR-21, miR-126, miR-146a and miR-222 levels at the above three different time was analyzed. One-step real-time quantitative polymerase chain reaction (RT-qPCR) was performed using a RT-qPCR system (T100TM Thermal Cycler, Bio-Rad Laboratories Inc., Berkeley, CA, USA) to assess plasma microRNA levels. A mixture of 100 ng total RNA extraction, 10 microL TaqMan master mix (ThermoFisher), 5.8 microL nuclease-free water, 0.2 microL universal probe library 21 (10 microM), 0.1 microL RNase inhibitor, self-constructed 1 microL forward primers and 1 microL reverse primers for miR-39, miR-126 and miR-146a, and 2 microL cDNA template were created on ice. All reactions were incubated in a 48-well plate at 95°C for 3 min, followed by 40 cycles of 95°C for 5 sec, 60°C for 10 sec and 72°C for 1 sec. Self-constructed forward and reverse primer sequences for primary C. elegans miR-39 (C-miR-39) as exogenous control. Human miR-126 (miR-126) and miR-146a (miR-146a) (Supplementary Table 1) were normalized by the exogenous control and were used to determine the microRNA levels expressions during the follow-up.

miRCURY LNA SYBR Green PCR kit (Qiagen) was used to determine human miR-21 (miR-21) and miR-222 (miR-222). A mixture of 4 microL 5X miRCURY RT SYBR Green Reaction Buffer, 2 microL 10X miRCURY RT Wnzyme Mix and 14 microL of 100 ng total RNA extraction in nuclease-free water was incubated in a 48-well plate at 42°C for 60 min and followed by 95°C to generate cDNA. A mixture containing 2 microL C-miR-39 (or miR-21/ or miR-222) primers purchased from Qiagen, 10 microL miRCURY SYBR Green Master Mix, 2 microL nuclease-free water and 6 microL 5X generated cDNA template was incubated at 95°C for 2 min, followed by 40 cycles of 95°C for 10 sec and 56°C for 60 sec. has-miR-21 and hsa-miR-222 were normalized by the C-miR-39 and were used to determine the microRNA levels expressions during the follow-up.

Determination of inflammatory activity 300 microL of serum was diluted by 1:2 ratios. Loaded 50 microL of prepared samples per well and calibrators in duplicate onto the assay plate (Multiplex Human Cytokine Panel 1, Boster Biological Technology, Pleasanton, CA, USA). Each well containing antibodies captured IL-1α, IL-1β, IL-6, IL-10, and TNFα. A mixture that contains biotinylated analyte specific antibodies is added after washing away any unbound protein. The biotinylated antibodies completed the sandwich for each specific arrayed analyte. After washing away unbound biotinylated antibody, streptavidin horseradish peroxidase (SHRP) is added. Following an additional wash, the amount of SHRP remaining on each location of the array is proportional to the amount of the above initially captured cytokines. The amount of conjugated enzyme on each location of the array is measured with the addition of a chemiluminescent substrate.

Statistical analysis Data are presented as mean (95% CI) or n (%). Differences of continuous and nominal parameters and between the two groups were estimated by student-t and chi-square tests, respectively. Repeated measurement ANOVA was conducted to analyze differences of continuous parameters measured at the three time points in each group. Pearson correlation was performed to find the relationship between physical fitness and miRNAs. A p value less than 0.05 was considered as statistical significance.

ELIGIBILITY:
Inclusion Criteria:

Primary

1.Community-indwelling individuals with age>=55 years, who lived adjacent to a community hospital were surveyed.

Secondary

1. Adults with mini-mental state examination (MMSE) score > 24
2. Negative lumbar spine as well as lower extremity degenerative joint disorder were recruited.

Exclusion Criteria:

1. unstable angina
2. unstable BP
3. severe aortic stenosis
4. inflammatory disease within recent 3 months
5. uncontrolled or severe cardiac dysrhythmias
6. uncompensated HF
7. embolic disease within recent 3 months
8. ST segment displacement>=2 mm at rest
9. uncontrolled diabetes
10. sarcopenia
11. Patients with absolute contraindications of exercise training (Pescatello LS, Arena R, Riebe D and Thompson PD. ACSM's guidelines for exercise testing and prescription. 9th ed. Philadelphia, PA.: Wolters Kluwer/Lippincott Williams & Wilkins; 2014.)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
walking steps per day (stp/d) | 24 weeks
  mean every day walking steps in a week measured by a wrist-worn smart watch
energy expenditure per day (Kcal/d) | 24 weeks
  mean every day energy consumption in a week estimated by a wrist-worn smart watch.
estimated maximum oxygen consumption (eVO2max) | Initial recruitment
  maximum energy consumption estimated from 2-min step numbers measured by an interactive voices and 3D depth imaging device.
estimated maximum oxygen consumption (eVO2max) | 8 weeks after recruitment
  maximum energy consumption estimated from 2-min step numbers measured by an interactive voices and 3D depth imaging device.
estimated maximum oxygen consumption (eVO2max) | 24 weeks after recruitment
  maximum energy consumption estimated from 2-min step numbers measured by an interactive voices and 3D depth imaging device.
Calf circumference (cm) | Initial recruitment
  Average maximum calf circumference of bilateral legs obtained by measuring tape.
Calf circumference (cm) | 8 weeks after recruitment
  Average maximum calf circumference of bilateral legs obtained by measuring tape.
Calf circumference (cm) | 24 weeks after recruitment
  Average maximum calf circumference of bilateral legs obtained by measuring tape.
5-time sit-to-stand duration (second) | Initial recruitment
  5-time sit-to-stand duration measured by an interactive voices and 3D depth imaging device.
5-time sit-to-stand duration (second) | 8 weeks after recruitment
  5-time sit-to-stand duration measured by an interactive voices and 3D depth imaging device.
5-time sit-to-stand duration (second) | 24 weeks after recruitment
  5-time sit-to-stand duration measured by an interactive voices and 3D depth imaging device.
Sit-and-reach distance (cm) | Initial recruitment
  Hand reaching distance while performing forward bending in a sitting position
Sit-and-reach distance (cm) | 8 weeks after recruitment
  Hand reaching distance while performing forward bending in a sitting position
Sit-and-reach distance (cm) | 24 weeks after recruitment
  Hand reaching distance while performing forward bending in a sitting position
Normalized total body water content (%) | Initial recruitment
  Total body water content obtained from bioimpedance measurement and was then normalized by body weight
Normalized total body water content (%) | 8 weeks after recruitment
  Total body water content obtained from bioimpedance measurement and was then normalized by body weight
Normalized total body water content (%) | 24 weeks after recruitment
  Total body water content obtained from bioimpedance measurement and was then normalized by body weight
Normalized total mineral content (%) | Initial recruitment
  Total body mineral content obtained from bioimpedance measurement and was then normalized by body weight.
Normalized total mineral content (%) | 8 weeks after recruitment
  Total body mineral content obtained from bioimpedance measurement and was then normalized by body weight.
Normalized total mineral content (%) | 24 weeks after recruitment
  Total body mineral content obtained from bioimpedance measurement and was then normalized by body weight.
Normalized total protein amount (%) | Initial recruitment
  Total body protein amount obtained from bioimpedance measurement and was then normalized by body weight.
Normalized total protein amount (%) | 8 weeks after recruitment
  Total body protein amount obtained from bioimpedance measurement and was then normalized by body weight.
Normalized total protein amount (%) | 24 weeks after recruitment
  Total body protein amount obtained from bioimpedance measurement and was then normalized by body weight.
Normalized body fat mass (%) | Initial recruitment
  Total body fat amount obtained from bioimpedance measurement and was then normalized by body weight.
Normalized body fat mass (%) | 8 weeks after recruitment
  Total body fat amount obtained from bioimpedance measurement and was then normalized by body weight.
Normalized body fat mass (%) | 24 weeks after recruitment
  Total body fat amount obtained from bioimpedance measurement and was then normalized by body weight.
Normalized skeletal mass to lean body mass percentage (%) | Initial recruitment
  Total skeletal mass obtained from bioimpedance measurement and was then normalized by lean body mass.
Normalized skeletal mass to lean body mass percentage (%) | 8 weeks after recruitment
  Total skeletal mass obtained from bioimpedance measurement and was then normalized by lean body mass.
Normalized skeletal mass to lean body mass percentage (%) | 24 weeks after recruitment
  Total skeletal mass obtained from bioimpedance measurement and was then normalized by lean body mass.
miR-21 (relative intensity) | Initial recruitment
  Ratio of human micro RNA 21 measured by real-time quantitative polymerase chain reaction compared to the level of microRNA 39 of C. elegans.
miR-21 (relative intensity) | 8 weeks after recruitment
  Ratio of human micro RNA 21 measured by real-time quantitative polymerase chain reaction compared to the level of microRNA 39 of C. elegans.
miR-21 (relative intensity) | 24 weeks after recruitment
  Ratio of human micro RNA 21 measured by real-time quantitative polymerase chain reaction compared to the level of microRNA 39 of C. elegans.
miR-126 (relative intensity) | Initial recruitment
  Ratio of human micro RNA 126 measured by real-time quantitative polymerase chain reaction compared to the level of microRNA 39 of C. elegans.
miR-126 (relative intensity) | 8 weeks after recruitment
  Ratio of human micro RNA 126 measured by real-time quantitative polymerase chain reaction compared to the level of microRNA 39 of C. elegans.
miR-126 (relative intensity) | 24 weeks after recruitment
  Ratio of human micro RNA 126 measured by real-time quantitative polymerase chain reaction compared to the level of microRNA 39 of C. elegans.
miR-146a (relative intensity) | Initial recruitment
  Ratio of human micro RNA 146a measured by real-time quantitative polymerase chain reaction compared to the level of microRNA 39 of C. elegans.
miR-146a (relative intensity) | 8 weeks after recruitment
  Ratio of human micro RNA 146a measured by real-time quantitative polymerase chain reaction compared to the level of microRNA 39 of C. elegans.
miR-146a (relative intensity) | 24 weeks after recruitment
  Ratio of human micro RNA 146a measured by real-time quantitative polymerase chain reaction compared to the level of microRNA 39 of C. elegans.
miR-222 (relative intensity) | Initial recruitment
  Ratio of human micro RNA 222 measured by real-time quantitative polymerase chain reaction compared to the level of microRNA 39 of C. elegans.
miR-222 (relative intensity) | 8 weeks after recruitment
  Ratio of human micro RNA 222 measured by real-time quantitative polymerase chain reaction compared to the level of microRNA 39 of C. elegans.
miR-222 (relative intensity) | 24 weeks after recruitment
  Ratio of human micro RNA 222 measured by real-time quantitative polymerase chain reaction compared to the level of microRNA 39 of C. elegans.
IL-1a (relative intensity) | Initial recruitment
  Ratio of IL-1a obtained from ELISA assay plate at each time point to the baseline level.
IL-1a (relative intensity) | 8 weeks after recruitment
  Ratio of IL-1a obtained from ELISA assay plate at each time point to the baseline level.
IL-1a (relative intensity) | 24 weeks after recruitment
  Ratio of IL-1a obtained from ELISA assay plate at each time point to the baseline level.
IL-1b (relative intensity) | Initial recruitment
  Ratio of IL-1b obtained from ELISA assay plate at each time point to the baseline level.
IL-1b (relative intensity) | 8 weeks after recruitment
  Ratio of IL-1b obtained from ELISA assay plate at each time point to the baseline level.
IL-1b (relative intensity) | 24 weeks after recruitment
  Ratio of IL-1b obtained from ELISA assay plate at each time point to the baseline level.
IL-6 (relative intensity) | Initial recruitment
  Ratio of IL-6 obtained from ELISA assay plate at each time point to the baseline level.
IL-6 (relative intensity) | 8 weeks after recruitment
  Ratio of IL-6 obtained from ELISA assay plate at each time point to the baseline level.
IL-6 (relative intensity) | 24 weeks after recruitment
  Ratio of IL-6 obtained from ELISA assay plate at each time point to the baseline level.
IL-10 (relative intensity) | Initial recruitment
  Ratio of IL-10 obtained from ELISA assay plate at each time point to the baseline level.
IL-10 (relative intensity) | 8 weeks after recruitment
  Ratio of IL-10 obtained from ELISA assay plate at each time point to the baseline level.
IL-10 (relative intensity) | 24 weeks after recruitment
  Ratio of IL-10 obtained from ELISA assay plate at each time point to the baseline level.
TNFa (relative intensity) | Initial recruitment
  Ratio of IL-10 obtained from ELISA assay plate at each time point to the baseline level.
TNFa (relative intensity) | 8 weeks after recruitment
  Ratio of IL-10 obtained from ELISA assay plate at each time point to the baseline level.
TNFa (relative intensity) | 24 weeks after recruitment
  Ratio of IL-10 obtained from ELISA assay plate at each time point to the baseline level.
Physical component score (PCS) | Initial recruitment
  Physical role function obtained from short form 36 questionnaire (SF-36) before and after exercise training. The SF-36 consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Physical component score (PCS) | 24 weeks after recruitment
  Physical role function obtained from short form 36 questionnaire (SF-36) before and after exercise training. The SF-36 consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Mental component score (MCS) | Initial recruitment
  Mental health score obtained from short form 36 questionnaire (SF-36) before and after exercise training. The SF-36 consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Mental component score (MCS) | 24 weeks after recruitment
  Mental health score obtained from short form 36 questionnaire (SF-36) before and after exercise training. The SF-36 consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chin Hsu, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Keelung Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No